CLINICAL TRIAL: NCT05473208
Title: "Effectiveness of Lumbar Assistive Exoskeleton in Nursing Home Caregivers: Randomized Control Trial"
Brief Title: Lumbar Assistive Exoskeletons in Caregiving
Acronym: ExoCare
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: Diputación Foral de Bizkaia (Unknown)
Responsible Party: Principal Investigator, Maialen Aiestaran, MsC, Principal Investigator, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ExoCare
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Healthy; Low Back Pain; Musculoskeletal Pain; Musculoskeletal Injury
Keywords: Low back pain; Exoskeleton; Caregiver; Nursing home; Musculoskeletal disease; Quality of life
MeSH Terms: conditions — Low Back Pain; Musculoskeletal Pain; Musculoskeletal Diseases | interventions — Exoskeleton Device

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators in charge of doing the statistical analysis and assessing the outcome measures (e.g., physical performance tests) will be blinded to group allocation. Due to the characteristics of the study (use of the exoskeleton during working hours) blinding of the participants is not possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants randomly assigned to control group will not wear an exoskeleton during working hours.
- Exoskeleton Group (Experimental): Participants randomly assigned to exoskeleton group will be given instructions and explanations on how to use/adjust/loosen the exoskeleton, and after a period of familiarisation, they will be wearing an exoskeleton during their working hours for a period of one year.
  Interventions: Device: Exoskeleton

INTERVENTIONS:
Device: Exoskeleton — Lumbar assistive exoskeleton evaluation
  Arms: Exoskeleton Group

SUMMARY:
A randomized control trial will be conducted, for evaluating the effectiveness of the implementation of a lower back assistive exoskeleton on the caregivers working in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* nursing home caregivers

Exclusion Criteria:

* pregnancy
* presence of condition that prevents from the use of a lumbar exoskeleton

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Pain Intensity at 3 months | At Baseline and at 3 months
  Average pain intensity during the last 7 days in a Numerical Rating Scale for pain ranging from 0 (complete absence of pain) to 10 (worst imaginable pain). This information will be collected for pain in the low back, neck, shoulders and wrists/hands
Change from baseline Pain Intensity at 6 months | At Baseline and at 6 months
  Average pain intensity during the last 7 days in a Numerical Rating Scale for pain ranging from 0 (complete absence of pain) to 10 (worst imaginable pain). This information will be collected for pain in the low back, neck, shoulders and wrists/hands
Change from baseline Pain Intensity at 9 months | At Baseline and at 9 months
  Average pain intensity during the last 7 days in a Numerical Rating Scale for pain ranging from 0 (complete absence of pain) to 10 (worst imaginable pain). This information will be collected for pain in the low back, neck, shoulders and wrists/hands
Change from baseline Pain Intensity at 12 months | At Baseline and at 12 months
  Average pain intensity during the last 7 days in a Numerical Rating Scale for pain ranging from 0 (complete absence of pain) to 10 (worst imaginable pain). This information will be collected for pain in the low back, neck, shoulders and wrists/hands

SECONDARY OUTCOMES:
Usability measured by System Usability Scale | Baseline, month 3, month 6, month 9, post intervention
  It is a simple scale of ten items that provides a subjective global vision of the usability of the evaluated exoskeleton on a scale of 1 to 5 (1 being strongly disagree and 5 strongly agree). Higher values mean the users found the device more usable.
User Satisfaction measured by Quebec User Evaluation of Satisfaction with Assistive Technology | Baseline, month 3, month 6, month 9, post intervention
  Scale to evaluate the satisfaction of the person during the use of the exoskeleton. It is made up of two subscales: the first considers eight aspects related to the support product (in this case, the exoskeleton); the second subscale evaluates four items regarding maintenance services during the use of the device. The scale goes from 1 (not satisfied at all) to 5 (very satisfied). Higher values mean that users are more satisfied.
Self-reported work ability by Work Ability Index | Baseline, month 3, month 6, month 9, post intervention
  It yields a continuous score ranging from 7 to 49 points, where higher scores indicate better work ability.
Borg's CR-10 scale for perceived physical exertion at work | Baseline, month 3, month 6, month 9, post intervention
  It measures perceived physical exertion while doing physical work in a scale ranging from 0 (nothing at all) to 10 (extremely strong).
Muscular resistance of the trunk muscles measured by the "Shirado-Ito" test | Baseline, month 3, month 6, month 9, post intervention
  It measures trunk muscle endurance based on the maximum time the participant is able to maintain a defined body position.
Discomfort measured by Body Part Discomfort Scale | Baseline, month 3, month 6, month 9, post intervention
  Survey of subjective symptoms that evaluates both the direct experience of discomfort of the person surveyed in different parts of the body, as well as the intensity of said discomfort on a scale of 0 to 10 (0 being no discomfort and 10 extremely high discomfort).
Absenteeism | Baseline, month 3, month 6, month 9, post intervention
  Days of absence from work will be collected from the official registry of the company and by the following question: "In total, how many days of work have you missed due to health reasons (injury, illness, medical consultation / treatment ...) during the last 12 weeks?". Possible answers will be: "0 days", "1-7 days", "8-30 days", "more than 30 days". In addition, number of days of absenteeism during the last 7 days (0-7) will be recorded.
Musculoskeletal disorders prevalence | Baseline, month 3, month 6, month 9, post intervention
  Prevalence of musculoskeletal injuries such as tendinopathies, unspecific low back pain
Prevalence of Side Effects | Baseline, month 3, month 6, month 9, post intervention
  Side effects secondary to the use of the exoskeleton such as: chafe, irritation, pressures.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez Larrad, PhD, Study Director — Professor
Locations (2):
- Spain (2):
  - IFAS/GUFE Centro Asistencial Leioa, Leioa, Bizkaia
  - IFAS/GUFE Centro Asistencial Elorrio, Elorrio, Vizcaya

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing under acceptable request